CLINICAL TRIAL: NCT05106478
Title: A Randomized Comparison of Pediatric® AuraGain in Supine, Moderate Lateral, and Extreme Lateral Positions in Terms of Clinical Performance and Fiber Optic Glottic
Brief Title: AuraGain Performance in Lateral Position
Acronym: AuraGainLMA
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Principal investigator, Assiut University
Other Study IDs: 17101416
Record Dates: First submitted 2021-10-09; First posted 2021-11-03 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Airway Complication of Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moderate lateral Group: Patients will be anesthetized using ® AuraGain airway that will be inserted lubricated with partially deflated cuff. After insertion, the cuff will be inflated with the recommended volume of air and operation will undergo while patient's neck in moderate lateral position.
  Interventions: Device: AuraGain
- Extreme lateral Group: Patients will be anesthetized using ® AuraGain airway that will be inserted lubricated with partially deflated cuff. After insertion, the cuff will be inflated with the recommended volume of air and operation will undergo while patient's neck in extreme lateral position.
  Interventions: Device: AuraGain

INTERVENTIONS:
Device: AuraGain — Ambu® AuraGain, a relatively novel supraglottic airway device, has been introduced recently. AuraGain has an inflatable cuff and a curved body.

SUMMARY:
To compare the clinical performance of AuraGain including insertion time and success rate at first attempt, fiberoptic bronchoscopic view, oropharyngeal leak pressure, the degree of ease of gastric tube insertion, and peri-operative adverse effects in young children in supine, moderate lateral and extreme lateral position.

DETAILED DESCRIPTION:
Ambu® AuraGain, a relatively novel supraglottic airway device, has been introduced recently. AuraGain has an inflatable cuff and a curved body. In addition, because the airway tube of AuraGain is wide, it can be used as a conduit for tracheal intubation. However, only a limited number of studies have been conducted on the performance of AuraGain in pediatric patients.

Changes in the position of the head and neck alter the shape of the pharynx leading to changes in the oropharyngeal leak pressure and the quality of ventilation through the LMA in both the adult and pediatric population. Having a large occiput and a relatively cephalically placed glottis, the ventilation in children is more compromised due to poor alignment of the pharyngeal-laryngeal axes during flexion of the head and neck. The hanging epiglottis covers the laryngeal inlet during flexion and the cuff of the LMA compresses the narrow laryngeal inlet both decreasing the delivered tidal volume. Different changes occur during extension and lateral rotation

Although the clinical performance of the AuraGain would be expected to be high, or at least non-inferior, to that of the widely used currently available SGAs, clinical trials are required to verify its performance in head and neck positions other than the neutral position (i.e flexion, extension and lateral rotation).

ELIGIBILITY:
Inclusion Criteria:

* Weight: 15-30 kg.
* Age: 2-9 years.
* Sex: both males and females.
* ASA physical status: 1-3.
* Operation: elective outpatient surgery in which airway management with a® AuraGain would be appropriate.

Exclusion Criteria:

* Active respiratory illness (cough, fever, rhinorrhea) on the day of anesthesia,
* Potentially difficult airway.
* Patients with history of neck, respiratory, or digestive tract pathology.
* Patients with gastroesophageal reflux, gastrointestinal stenosis, or stricture.

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: - children scheduled for elective outpatient surgery in which airway management with a® AuraGain would be appropriate.
Sampling Method: Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | Intraoperative from 1 minute after insertion of the device as a baseline to 60 minutes after insertion of the device
  Airway leak pressure will be determined by closing the adjustable expiratory pressure-limiting (APL) valve and setting the fresh gas flow rate to 3 L/min. The airway pressure at which an audible leak in the mouth is heard is recorded as the "leak Pressure".

SECONDARY OUTCOMES:
Ventilation score (grade 0, 1, 2 or 3), | Intraoperative from 1 minute after insertion of the device as baseline to 60 minutes after insertion of the device
  the ventilation score which is scored from 0 to 3 based on three criteria: no leakage with an airway pressure of 15 cm H2O, bilateral chest excursions with a peak inspiratory pressure of 20 cm of H2O, and a square wave capnogram, with each item scoring 0 or 1 point . Thus, if all three criteria are satisfied, the ventilation score is 3.
Fiberoptic glottic view Score | Intraoperative from 1 minute after insertion of the device to 60 minutes after insertion of the device.
  The fiberoptic images will be graded with a score from 1 to 5, which has been defined and proposed previously (20, 21); (grade 1-only larynx seen; grade 2-larynx and epiglottis posterior surface seen; grade 3-larynx and epiglottis tip of anterior surface seen, <50%visual obstruction of epiglottis to larynx; grade 4-epiglottis down folded and its anterior surface seen, >50%visual obstruction of epiglottis to larynx; and grade 5-epiglottis down folded and larynx cannot be seen directly). The images will be taken in the neutral position and in mid and extreme laterally rotated neck positions.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assiut University
Locations (1):
- Hala Abdel-Ghaffar, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No